CLINICAL TRIAL: NCT05169463
Title: NETTUNIT - Italy-Tunisia Cross-border Environmental network_1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Stefania La Grutta, MD, Research Director, Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: 03/2021_1
Record Dates: First submitted 2021-11-16; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Respiratory Disease; Cardiovascular Diseases
MeSH Terms: conditions — Respiration Disorders; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective, case-crossover study aiming to use environmental pollutant data for assessing the associated risk of visiting the emergency room (ER) for respiratory or cardiovascular problems in the territory of the Caltanissetta Provincial Health Authority (Italy). All the ER visits for respiratory and/or cardiovascular disorders in the hospital of Gela (Italy) and Niscemi (Italy) from 2010 to 2019 will be considered.

ELIGIBILITY:
Inclusion Criteria:

* All emergency room visits for respiratory or cardiovascular problems at the hospital of Gela (Italy) and Niscemi (Italy), from 2010 to 2019.

Exclusion Criteria:

* Emergency room visits for other diseases.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All emergency room visits for respiratory or cardiovascular problems at the hospital of Gela (Italy) and Niscemi (Italy), from 2010 to 2019.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-03-03 (Estimated); Study Completion 2023-03-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of emergency room visit for respiratory diseases (binary outcome) | From year 2010 to year 2019
  Dates of emergency room visits (case days) for respiratory diseases will be retrieved and linked to air pollution data. For each case day, the binary outcome will be equal to 1. For the two control days (7 days before/after the case day), the binary outcome will be equal to 0.
Occurrence of emergency room visit for cardiovascular diseases (binary outcome) | From year 2010 to year 2019
  Dates of emergency room visits (case days) for cardiovascular diseases will be retrieved and linked to air pollution data. For each case day, the binary outcome will be equal to 1. For the two control days (7 days before/after the case day), the binary outcome will be equal to 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Palermo, Italy